CLINICAL TRIAL: NCT00264862
Title: Use of DynaCT in Endovascular Treatment of Abdominal Aortic Aneurysm. Evaluation of Image Quality.
Brief Title: DynaCT Imaging in EVAR: Comparing Clinical Benefit of DynaCT to Multidetector CT as the Current Gold Standard.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FOR2008_1
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: DynaCT

SUMMARY:
The aim of this study is to evaluate a new way to create CT-like images during intra-operative procedures. We want to prove that the quality and information received from DynaCT is satisfactory in implementing stent-graft in abdominal aortic aneurysm.

DETAILED DESCRIPTION:
The study will compare images from the new modality (DynaCT) with the present modality (Multi detectorCT). We make three different set of images from each modality.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65,
* Satisfactory renal function

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-12; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Evidence og clinical benefit of new imaging functionality. | 3 days (pluss or minus 3 days).

CONTACTS AND LOCATIONS:
Overall Officials: Kari R Eide, MS, Principal Investigator — NTNU/St.Olavs Hospital; Olav Haraldseth, PhD MD, Study Chair — National Taiwan Normal University
Locations (1):
- St. Olavs Hosptial, Trondheim, Norway

REFERENCES:
- [Result] Eide KR, Odegard A, Myhre HO, Lydersen S, Hatlinghus S, Haraldseth O. DynaCT during EVAR--a comparison with multidetector CT. Eur J Vasc Endovasc Surg. 2009 Jan;37(1):23-30. doi: 10.1016/j.ejvs.2008.09.017. Epub 2008 Nov 17. PMID 19010697